CLINICAL TRIAL: NCT02292407
Title: AND Precise! : Axillary Lymph Node Dissection and No Drain With the PRECISE Instrument
Brief Title: Prospective Pilot Study ANDPrecise
Acronym: ANDPrecise
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N12PRE
Record Dates: First submitted 2014-10-27; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LigaSure Precise instrument (Experimental): ALND with use of LigaSure Precise instrument, closure of dead space, omission of a postoperative drain.
  Interventions: Device: LigaSure Precise instrument

INTERVENTIONS:
Device: LigaSure Precise instrument — LigaSure Precise instrument is used during Axillary Lymph Node Dissection Technique: Dead space closure Technique: Omission of postoperative drain

SUMMARY:
This study aims at providing first evidence that axillary clearance by using an operation technique including the precise LigaSure instrument and closure of dead space of the axilla will result in an operation were a drain is not necessary and the need for seroma evacuation after surgery is very limited.

DETAILED DESCRIPTION:
Axillary clearance in breast cancer is usually performed by using a drain to prevent seroma formation and to support obliteration of the dead space in the axillary carry out. The hypothesis made in this protocol is that axillary clearance by using an operation technique including the use of the precise LigaSure instrument and closure of dead space can be done without using a postoperative drain.

The AND PRECISE PROTOCOL aims at providing first evidence that axillary clearance by using an operation technique including the precise LigaSure instrument and closure of dead space of the axilla will result in an operation were a drain is not necessary and the need for seroma evacuation after surgery is very limited Patients undergoing axillary clearance necessary for achieving reasonable control in invasive breast cancer and participating in the AND PRECISE protocol will undergo the operation by using a technique including the use of the precise LigaSure instrument and closure of dead space. Postoperatively, the numbers of seroma punctions and the amount of seroma will be recorded prospectively. Patients will be asked to record on a daily basis their experience of pain by a visual analog scale of pain.

The main study parameter is the percent of cases which successfully did not need seroma punctions after the intervention.

Potential disadvantages for the patient are risk for more seroma formation and discomfort. Patients will be asked to record on a daily basis their experience of pain by a visual analog scale of pain.

ELIGIBILITY:
Inclusion Criteria:

* Indications for axillary clearance can be a tumor positive sentinel node or tumor positive lymph nodes proven by ultrasound or fine needle aspiration cytology.
* For this pilot, only patients undergoing breast conserving surgery are eligible.
* Axillary clearance can be performed after previous sentinel node procedure, at the same operation, and after neo-adjuvant chemo therapy, and as secondary procedure in case of axillary relapse after previous treatment for breast cancer.

Exclusion Criteria:

* Patients undergoing a modified radical mastectomy including an axillary clearance.
* Preoperative preexisting seroma.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of seroma evacuations per patient | within 3 months after surgery

SECONDARY OUTCOMES:
Number of wound infections per patient | within 3 months after surgery
Number of hematomas per patient | within 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emiel Rutgers, MD, PhD, Principal Investigator — Netherlands Cancer Institute - Antoni van Leeuwenhoek
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, Netherlands

REFERENCES:
- [Background] van Bemmel AJ, van de Velde CJ, Schmitz RF, Liefers GJ. Prevention of seroma formation after axillary dissection in breast cancer: a systematic review. Eur J Surg Oncol. 2011 Oct;37(10):829-35. doi: 10.1016/j.ejso.2011.04.012. Epub 2011 Aug 17. PMID 21849243
- [Background] Baas-Vrancken Peeters MJ, Kluit AB, Merkus JW, Breslau PJ. Short versus long-term postoperative drainage of the axilla after axillary lymph node dissection. A prospective randomized study. Breast Cancer Res Treat. 2005 Oct;93(3):271-5. doi: 10.1007/s10549-005-5348-7. PMID 16172795
- [Background] Classe JM, Berchery D, Campion L, Pioud R, Dravet F, Robard S. Randomized clinical trial comparing axillary padding with closed suction drainage for the axillary wound after lymphadenectomy for breast cancer. Br J Surg. 2006 Jul;93(7):820-4. doi: 10.1002/bjs.5433. PMID 16775817
- [Background] Ostapoff KT, Euhus D, Xie XJ, Rao M, Moldrem A, Rao R. Axillary lymph node dissection for breast cancer utilizing Harmonic Focus(R). World J Surg Oncol. 2011 Aug 15;9:90. doi: 10.1186/1477-7819-9-90. PMID 21843361
- [Background] Gong Y, Xu J, Shao J, Cheng H, Wu X, Zhao D, Xiong B. Prevention of seroma formation after mastectomy and axillary dissection by lymph vessel ligation and dead space closure: a randomized trial. Am J Surg. 2010 Sep;200(3):352-6. doi: 10.1016/j.amjsurg.2009.10.013. Epub 2010 Apr 20. PMID 20409509